CLINICAL TRIAL: NCT01729533
Title: The Benefits of Intracytoplasmic Morphologically Selected Sperm Injection (IMSI) in Couples With Unexplained Infertility
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Sapientiae Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMSI_unexplained infertility
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Pregnancy
Keywords: ICSI; IMSI; Pregnancy; Sperm morphology; Unexplained infertility
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICSI (Active Comparator): In this arm, patients will be provided with standard intracytoplasmic sperm injection (ICSI), in which sperm selection is performed under an overall magnification of x400.
  Interventions: Other: ICSI
- IMSI (Experimental): In this arm, patients will be provided with a modified intracytoplasmic sperm injection (ICSI) procedure, the IMSI, in which sperm selection is performed under an overall magnification of x6600.
  Interventions: Other: IMSI

INTERVENTIONS:
Other: ICSI — ICSI Sperm selection in the ICSI group is analyzed under a magnification of 400x using an inverted microscope. ICSI is performed in a micro-injection dish prepared with 4 µL droplets of buffered medium and covered with paraffin oil on a heated stage at 37.0 ± 0.5°C of an inverted microscope.
  Other Names: Intracytoplasmic sperm injection
  Arms: ICSI
Other: IMSI — Sperm selection in the IMSI group is analyzed at high magnification using an inverted microscope equipped with high-power differential interference contrast optics. The total calculated magnification is x6.600. The sperm cells exhibiting normally shaped nuclei ([1] smooth, [2] symmetric, and [3] oval configuration) and [4] normal nuclear chromatin content (if it contained no more than one vacuole, which occupies <4% of the nuclear area) are selected for injection.
  Other Names: Intracytoplasmic morphologically selected sperm injection
  Arms: IMSI

SUMMARY:
The (motile sperm organelle morphology examination) MSOME allows the detection of sperm vacuoles that seems to be related to sperm DNA damage.

The investigators hypothesized that couples with unexplained infertility could benefit from the injection of spermatozoa selected under high-magnification (x6600)

DETAILED DESCRIPTION:
When routine infertility workup yields normal results in both partners, the couple is defined as suffering from unexplained infertility. These couples present normal semen analysis.

It has been reported that even infertile patients with normozoospermic parameters can have higher values of DNA damage than fertile controls.

It has been proposed that the use of ''invisible damaged'' spermatozoa could result in fertilization failure, impaired normal embryo development, reduced implantation and pregnancy rates.

The motile sperm organelle morphology examination (MSOME) allows the detection of sperm vacuoles that seems to be related to sperm DNA damage.

The investigators hypothesized that couples with unexplained infertility could benefit from the injection of spermatozoa selected under high-magnification (x6600)

ELIGIBILITY:
Inclusion Criteria:

* Women of good physical and mental health
* Undergoing assisted reproduction as a result of unexplained infertility
* Women with regular menstrual cycles of 25-35 days
* Women with normal basal follicle stimulating hormone (FSH) and luteinizing hormone (LH) levels
* Women with body mass index (BMI) less than 30 kg/m2
* Women with both ovaries and intact uterus

Exclusion Criteria:

* Men with abnormal semen parameters according to the 2010 WHO values
* Women with polycystic ovaries
* Women with endometriosis
* Women with gynaecological/medical disorders
* Women or men with a positive result for sexually transmitted diseases
* Women who had received hormone therapy for at least 60 days preceding the study

Max Age: 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 1 month
  Number of pregnancies divided by the number of cycles with embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Sapientiae Institute, São Paulo, São Paulo, Brazil